CLINICAL TRIAL: NCT03810404
Title: The Effect of Acute Sodium Bicarbonate Supplementation on Buffering Potential Kinetics, Physical Capacity and Discipline-Specific Performance
Brief Title: Acute Sodium Bicarbonate Supplementation in Athletes
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Principal Investigator, Poznan University of Physical Education
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ULS00006
Record Dates: First submitted 2019-01-14; First posted 2019-01-18 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Supplementation; Sport
Keywords: Sports nutrition; Sodium bicarbonate; Physical capacity; Exercise performance; Buffering potential; Biochemical markers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium bicarbonate supplementation (Experimental): Group taking oral SB supplementation in a different-dose regimen.
  Interventions: Dietary Supplement: Sodium bicarbonate supplementation
- Placebo treatment (Placebo Comparator): Group taking oral supplementation with placebo (NaCl).
  Interventions: Dietary Supplement: Placebo treatment

INTERVENTIONS:
Dietary Supplement: Sodium bicarbonate supplementation — Interventions:
  The experimental procedure for each athlete included an acute SB supplementation in a different-dose regimen in order to assess whether the dose affects the actual physical and exercise capacity (doses: 0.15-, 0.25-, 0.35- and 0.50 g/kgFFM (0.12-, 0.20-, 0.28- and 0.40 g/kgBM), respectively). SB (Alkala, SANUM, Poland) will be administered as dissolved form in a 750 ml of fluid (water + fruit juice). On testing days the SB will be taken before physical and exercise capacity tests session.
  Between the SB and PLA or a PLA and SB treatments, a minimum 7-day washout period will be introduced.
  Arms: Sodium bicarbonate supplementation
Dietary Supplement: Placebo treatment — Interventions:
  The experimental procedure for each athlete will be included an PLA supplementation. Placebo will be administered in a form of 750 ml of fluid (water + fruit juice). On testing days the PLA will be taken before physical and exercise capacity tests session.
  Between the PLA and SB or a SB and PLA treatments, a minimum 7-day washout period will be introduced.
  Arms: Placebo treatment

SUMMARY:
The purpose of this study is to verify the effect of acute sodium bicarbonate (SB) and placebo (PLA) supplementation on buffering potential kinetics, physical capacity, discipline-specific performance as well as concentration of diagnostically significant blood biochemical indices in athletes, in a randomised, double-blind, placebo-controlled crossover trial.

DETAILED DESCRIPTION:
Effective muscle work is conditioned by maintaining the proper range of muscles pH, regulated by buffering systems, in which the main role is played by bicarbonates (HCO3-). For this reason, sodium bicarbonate (SB) is often proposed as an ergogenic agent, especially during high-intensity efforts. Until now the major limitation to SB supplementation has been the gastrointestinal (GI) side effects. There is also a lack of data of the individual SB-induced changes of buffering potential kinetics and its actual connection with physical capacity and discipline-specific performance. Therefore, this study aims to examine the effect of acute, different-dose SB ingestion on buffering potential kinetics, physical capacity, discipline-specific performance as well as changes of diagnostically significant blood biochemical indices concentration in athletes, in a randomised, double-blind, placebo-controlled crossover trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* a current medical clearance to practice sports,
* training experience: at least 2 years,
* minimum of 4 workout sessions (in the discipline covered by the study) a week.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-01-20 (Estimated)

PRIMARY OUTCOMES:
Changes in anaerobic capacity after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  The Wingate cycling test carried out at baseline, and after SB and PLA supplementation
Changes in discipline-specific exercise capacity after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  The discipline-specific exercise capacity tests carried out at baseline, and after SB and PLA supplementation
Changes of bicarbonate concentration in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Bicarbonate (HCO3-) [mmol/L] concentration analysis in blood carried out at baseline, and after SB and PLA supplementation
Changes of base excess concentration in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Base excess [mmol/L] concentration analysis in blood carried out at baseline, and after SB and PLA supplementation

SECONDARY OUTCOMES:
Changes of pH in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Blood pH (pH units) analysis carried out at baseline, and after SB and PLA supplementation
Changes of lactate concentration in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Lactate [mmol/L] concentration analysis carried out at baseline, and after SB and PLA supplementation
Changes of pyruvate concentration in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Pyruvate [mmol/L] concentration analysis carried out at baseline, and after SB and PLA supplementation
Changes in blood glucose concentration after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Glucose [g/dl] concentration analysis carried out at baseline, and after SB and PLA supplementation
Changes in hemoglobin concentration after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Hemoglobin (Hb) [g/dl] concentration analysis carried out at baseline, and after SB and PLA supplementation
Changes of blood cells concentration in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Blood cells [mln/mm³] concentration analysis carried out at baseline, and after SB and PLA supplementation
Changes of creatine kinase activity in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Creatine kinase [U/L] activity analysis carried out at baseline, and after SB and PLA supplementation
Changes of lactate dehydrogenase activity in blood after sodium bicarbonate supplementation and placebo treatment | Baseline and during 1 day of acute SB and PLA supplementation
  Lactate dehydrogenase [U/L] activity analysis carried out at baseline, and after SB and PLA supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Durkalec-Michalski, Prof., PhD, Principal Investigator — Department of Sports Dietetics, Poznan University of Physical Education
Locations (1):
- Department of Sports Dietetics, Poznan University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level of recorded indicators, without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.